CLINICAL TRIAL: NCT05331170
Title: Epigenetic Mechanism Reprogramming Mucosal Anti-viral Immunity in Allergic Asthma VIRAL MUCOSAL REPROGRAMMING
Brief Title: Viral Mucosal Reprogramming
Acronym: VMR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: U01-UWM-01; 19-0240 (Other: UTMB Record ID)
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Asthma; Allergic Rhinitis; Cat Allergy; Healthy
Keywords: Asthma; Allergy; Allergic; Rhinitis; Airway; Cat dander; Respiratory
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Hypersensitivity; Rhinitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy (Active Comparator): Subjects without asthma, COPD, rhinitis and with negative allergen test
  Interventions: Biological: Research Grade RG-RV
- Allergic Rhinitis (Active Comparator): Subjects without asthma, COPD and with positive allergen test
  Interventions: Biological: Research Grade RG-RV
- Allergic Ashthma (Active Comparator): Subjects with asthma and positive allergen test
  Interventions: Biological: Research Grade RG-RV

INTERVENTIONS:
Biological: Research Grade RG-RV — Exploration of the effects of RV inoculation on human airway mucosal programming in vivo

SUMMARY:
This is a mechanistic, controlled, open-label, single-site study to evaluate the effects of RG-RV16 inoculation on airway mucosal gene expression and airway remodeling in 25 healthy controls (HC), in 25 allergic rhinitis subjects (AR) with cat dander allergy, and in 25 allergic asthmatic subjects (AA) with cat dander allergy. Three groups (HC, AR, and AA) will undergo screening to establish clinical history, will undergo pulmonary function testing (spirometry), and will have blood drawn for clinical characterization (IgE, , ImmunoCAP, CBC and differential), and for assessing the presence of existing neutralizing antibody against RV16. Only those who meet criteria will be permitted to continue into the interventional and run-out phases of the study.

ELIGIBILITY:
Inclusion Criteria:

Healthy Normal Control Group

1. Subject must be able to understand and provide informed consent
2. Age: 18-60 inclusive
3. Sex: M or F
4. No history of asthma, COPD, rhinitis, or other clinically important respiratory disease
5. Non-smoker, or ex-smoker with <10 pack years, at least 5 years remote.
6. No history of diabetes or cardiovascular disease
7. Negative ImmunoCAP test to regionally relevant allergen panel obtained at Screening. Alternatively, documented history of a negative skin test or negative specific IgE obtained within the past 12 months.

Allergic Rhinitis Group

1. Subject must be able to understand and provide informed consent
2. Age: 18-60 inclusive
3. Sex: M or F
4. No history of asthma, COPD, or other clinically important respiratory disease
5. Non-smoker, or ex-smoker with <10 pack years, at least 5 years remote
6. No history of diabetes or cardiovascular disease
7. History of rhinitis, physician diagnosed, plus one of the following criteria within the past 12 months
8. Seasonal or perennial nasal congestion or sneezing
9. Seasonal or perennial conjunctival infection or watering
10. No evidence of airway obstruction (FEV1:FVC ≥ lower limit of normal)
11. Positive ImmunoCAP test to cat. Documented history at any time of a positive skin test or a specific IgE measure at least Level 2 reactivity will meet this criterion. Subjects must have cat in home, have regular exposure to cat dander, or live in a home where a cat has lived within the past 6 months.

Allergic Asthma Group

Inclusion Criteria

1. Subject must be able to understand and provide informed consent
2. Age: 18-60 inclusive
3. Sex: M or F
4. No history of COPD or other clinically important respiratory disease other than asthma
5. Non-smoker, or ex-smoker with <10 pack years, at least 5 years remote
6. No history of diabetes or cardiovascular disease
7. History of mild-moderate asthma, physician diagnosed, plus one of the following criteria within the past 12 months

   1. Airway obstruction (FEV1: FVC <0.6) that is significantly (at least 12% change from baseline, ATS criteria) reversible after 4 puffs of albuterol (obtained at Screening Visit or documented historical testing performed with the past 12 months)
   2. Requiring ICS for control of asthma for at least 30 days within the past 12 months
8. Positive ImmunoCAP test to cat dander. Documented history at any time of a positive skin test or a specific IgE measure at least Level 2 reactivity will meet this criteria. Subjects must have cat in home, have regular exposure to cat dander, or live in a home where a cat has lived within the past 6 months.
9. Results of the CBC do not show clinically important abnormalities

Exclusion Criteria:

Healthy Group Normal Group

1. Inability or unwillingness of a participant to comply with study protocol
2. Currently taking inhaled corticosteroids, leukotriene modifier, or antihistamines for respiratory disease.
3. Neutralizing Ab to RV16 greater than or equal to 1:8
4. Pregnant or breastfeeding women or a woman who has a planned pregnancy during the course of the study. Menstruating females must have a negative pregnancy test at the screening visit. Pregnancy testing may be conducted prior to procedures as well at various times in the study.
5. Subjects with household or close contacts who are pregnant or planning a pregnancy during the main subject's participation, who have chronic respiratory disease, who are children under the age of 2 years, or who are adults over 60 years of age or are Immunosuppressed e.g. post-chemotherapy, HIV).
6. Subjects who provide healthcare services or work with elderly or children (e.g. daycare provider, senior citizen care giver).

Allergic Rhinitis Group

1. Inability or unwillingness of a participant to comply with study protocol
2. Currently using inhaled steroids, or oral montelukast for respiratory disease
3. Neutralizing Ab to RV16 greater than or equal to 1:8
4. Pregnant or breastfeeding women or a woman who has a planned pregnancy during the course of the study. Menstruating females must have a negative pregnancy test at screening visit. Pregnancy testing may be conducted prior to procedures as well at various times in the study.
5. Subjects with household or close contacts who are pregnant or planning a pregnancy during the main subject's participation, who have chronic respiratory disease, who are children under the age of 2 years, or who are adults over 60 years of age or are Immunosuppressed e.g. post-chemotherapy, HIV) .
6. Subjects who provide healthcare services or work with elderly or children (e.g. daycare provider, senior citizen care giver).
7. Subjects who have received immunosuppressive treatment within the last 12 months
8. BMI is greater than 35
9. History of symptoms consistent with a viral URI within the past 21 days
10. Results of the CBC do not show clinically important abnormalities
11. Family history or medical history of liver disease or bleeding disorders
12. Have not received systemic corticosteroids for 3months prior to Screening
13. Antiplatelet agents other than aspirin
14. Subjects who have a positive COVID-19 test will be excluded for 8 weeks

Allergic Asthma Group

1. Inability or unwillingness of a participant to comply with study protocol
2. Currently taking medications for respiratory diseases other than ICS, montelukast, or rescue albuterol or LABAs.
3. Neutralizing Ab to RV16 greater than or equal to 1:8
4. FEV1: FVC ratio less than 0.6, or FEV1 less than 60% predicted
5. Recent (<30 days) exacerbation of asthma requiring systemic corticosteroids
6. ICS greater than fluticasone 500 mcg/day or its equivalent (GINA 2019 table) at screening.
7. Pregnant or breastfeeding women or a woman who has a planned pregnancy during the course of the study. Menstruating females must have a negative pregnancy test at screening. Pregnancy testing may be conducted prior to procedures as well at various times in the study.
8. Subjects with household or close contacts who are pregnant or planning a pregnancy during the main subject's participation, who have chronic respiratory disease, who are children under the age of 2 years, or who are adults over 60 years of age or are Immunosuppressed e.g. post-chemotherapy, HIV) .
9. Subjects who provide healthcare services or work with elderly or children (e.g. daycare provider, senior citizen care giver).
10. Subjects who have received immunosuppressive treatment within the last 12 months
11. BMI is greater than 35
12. History of symptoms consistent with a viral URI within the past 21 days
13. Family history or medical history of liver disease or bleeding disorders
14. Have not received systemic corticosteroids for 3 months prior to Screening
15. Have an ACT score >19 at the time of enrollment.
16. Antiplatelet agents other than aspirin
17. Subjects who have a positive COVID-19 test will be excluded for 8 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
ZEB-1 Expression | Immediate
  Q-PCR
Type III Interferon | Immediate
  Q-RT-PCR
PD-L1 Expression | Immediate
  Q-RT-PCR
RV16 Viral Titer | 48 hours after inoculation
  Plaque Assays

SECONDARY OUTCOMES:
CD8 T cells in bronchoalveolar lavage fluid | Immediate and 48hrs post RV16 inoculation
  Proportion and number of CD8+ T cells
Airway Remodeling | Immediate and 48 hrs post RV16 inoculation
  Lamina reticularis thickness
URI Cold Symptoms | Immediate and up to 7 days following inoculation
  WURSS21 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: William J. Calhoun, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States